CLINICAL TRIAL: NCT00001631
Title: Study of Myocardial Perfusion by MRI
Brief Title: Study of Blood Flow in Heart Muscle
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970177; 97-H-0177
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-01

CONDITIONS: Coronary Disease; Healthy; Hypertrophic Cardiomyopathy; Myocardial Ischemia
Keywords: Gadolinium; Ischemia; Coronary Artery Disease; Hypertrophic Cardiomyopathy; Dipyridamole
MeSH Terms: conditions — Coronary Disease; Cardiomyopathy, Hypertrophic; Myocardial Ischemia; Ischemia; Coronary Artery Disease | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: Magnetic resonance imaging

SUMMARY:
Blood flows to areas of the heart providing oxygen and fuel to the pumping muscle. Occasionally the arteries providing the fuel can become blocked. This occurs in coronary artery disease.

Magnetic resonance imaging (MRI) can be used to evaluate the blood flow to different areas of the heart muscle. In this study magnetic resonance imaging will be compared to other diagnostic tests (radionucleotide perfusion studies) capable of measuring blood flow to heart muscle.

DETAILED DESCRIPTION:
In this pilot study, magnetic resonance imaging (MRI) of myocardial enhancement during first passage of intravenously injected gadolinium contrast will be used to evaluate regional myocardial perfusion in patients with known or suspected coronary artery disease and hypertrophic cardiomyopathy. The MRI results will be compared with conventional radionuclide perfusion studies (ex. dipyridamole thallium). A clinically defined normal group will also be studied without radionuclide correlation.

ELIGIBILITY:
INCLUSION CRITERIA:

Ages 18 to 80.

Either sex.

Capable of giving informed consent.

Group 1: Outpatients with known or suspected coronary artery disease with clinical indication for radionuclide perfusion imaging.

Group 2: Patients with non-obstructive hypertrophic cardiomyopathy with clinical indication for radionuclide perfusion imaging.

Group 3: Normal volunteers.

Positive stress thallium or stress sestamibi (i.e., exercise, adenosine, dobutamine or dypiridamole) at the NIH.

EXCLUSION CRITERIA:

Pregnancy.

Unstable angina.

Uncontrolled hypertension (SBP greater than 185, DBP greater than 105).

Recent myocardial infarction (less than 5 days).

2nd or 3rd degree heart block by ECG.

Asthma, emphysema, renal failure, acute medical illness (fever, pneumonia, etc.) or anemia (hct less than 30).

Cardiac pacemaker or implantable defibrillator, aneurysm clip, neural stimulator, any type of ear implant, metal in your eye, any implanted device (i.e. insulin pump, drug infusion device) or any metallic foreign body, shrapnel, or bullet.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 249
Dates: Start 1997-08; Study Completion 2003-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Wilke N, Simm C, Zhang J, Ellermann J, Ya X, Merkle H, Path G, Ludemann H, Bache RJ, Ugurbil K. Contrast-enhanced first pass myocardial perfusion imaging: correlation between myocardial blood flow in dogs at rest and during hyperemia. Magn Reson Med. 1993 Apr;29(4):485-97. doi: 10.1002/mrm.1910290410. PMID 8464365
- [Background] Matheijssen NA, Louwerenburg HW, van Rugge FP, Arens RP, Kauer B, de Roos A, van der Wall EE. Comparison of ultrafast dipyridamole magnetic resonance imaging with dipyridamole SestaMIBI SPECT for detection of perfusion abnormalities in patients with one-vessel coronary artery disease: assessment by quantitative model fitting. Magn Reson Med. 1996 Feb;35(2):221-8. doi: 10.1002/mrm.1910350214. PMID 8622587
- [Background] Zaman M, Hashmi R, Niaz K, Ahmad A, Kamal S. Safety of pharmacological (intravenous dipyridamole) stress for Thallium-201 perfusion imaging in patients with coronary artery disease unable to exercise. J Pak Med Assoc. 1994 Oct;44(10):237-9. PMID 7815687